CLINICAL TRIAL: NCT04992871
Title: Swiss Cerebral Palsy Registry
Acronym: Swiss-CP-Reg
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Schweizerische Stiftung für das cerebral gelähmte Kind (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-00873
Record Dates: First submitted 2021-07-22; First posted 2021-08-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Children, adolescents and adults diagnosed with cerebral palsy who are born, treated or living in Switzerland

SUMMARY:
The Swiss-CP-Reg is a national patient registry that collects information on diagnosis, symptoms, treatment and follow-up of patients with cerebral palsy (CP) in Switzerland. It was first implemented in 2017 in the paediatric clinics in Basel, Bellinzona, Bern, Geneva, Lausanne, St. Gallen and Zurich. It is currently extended to all Swiss clinics and medical practices and adults will be invited to join the register in the coming years. The registry provides data for national and international monitoring and research. It supports research on CP in Switzerland and the exchange of knowledge between clinicians, researchers and therapists, with the goal to improve the treatment of children and adults with CP and optimizing their health and quality of life.

DETAILED DESCRIPTION:
Background: Cerebral palsy (CP) refers to chronic movement and postural disorders. It results from a non-progressive lesion or brain malformation that occurs during the prenatal, perinatal, or postnatal period (e.g. ischemic lesions of the neonatal brain or genetic predispositions leading to brain malformation). Besides motor dysfunction, persons with CP suffer from a wide variety of comorbidities, such as epilepsy, speech, hearing or vision disorders, cognitive dysfunction, behavioral disorders, and secondary musculoskeletal problems.

CP is the most common cause of physical disability in children in Switzerland and it is important that the investigators gain a better understanding of its prevalence, risk factors, current clinical profile and the needs of those affected and their families.

The cantonal Ethics Committee of Bern approved the Swiss-CP-Reg project (project ID: 2017-00873, observational study, risk category A).

Objectives: The overall objective of the Swiss-CP-Reg is to improve future care and thus well-being of CP individuals. The development of a national registry for the collection of representative, complete and longitudinal data from children, adolescents and adults with CP in Switzerland serves to achieve this goal.

Primary objectives of the Swiss-CP-Reg projects:

1. Establish a representative population-based Swiss cohort of children, adolescents and adults with CP
2. Provide epidemiological data to investigate the incidence, prevalence, risk factors, spectrum of diagnosis, survival rates and mortality
3. Provide a platform for clinical research:

   * Answer questions in the following areas: health, health care, education, social aspects and quality of life
   * Offer a resource to recruit patients for nested observational and intervention studies
4. Provide a platform for communication:

   * Promote the exchange of knowledge between clinics, researchers, therapists and national and cantonal health authorities
   * Facilitate international collaborations, in particular with the "Surveillance of Cerebral Palsy of Europe" (SCPE), and benchmarking of used therapeutic approaches with international partners

Inclusion/exclusion criteria: all children, adolescents and adults diagnosed with CP who are born, treated or living in Switzerland. The SCPE decision tree is used for inclusion/exclusion. Patients with pure muscular hypotonia, neurometabolic diseases (e.g. neuronal storage diseases, leukodystrophies) and other progressive neurological diseases (e.g. spinocerebellar ataxias, hereditary spastic paraplegia, Rett syndrome, epileptic encephalopathy) are excluded.

Procedure: After a CP diagnosis of a child, the treating physician informs the family during a consultation in a clinic or practice in writing and orally about the Swiss-CP-Reg. Families who wish to participate sign the consent form and the children are registered in the Swiss-CP-Reg. If families do not wish to participate, only a minimal anonymous data set is recorded.

The following data will be collected:

* Medical data
* Data from questionnaires for patients and families
* Data from links to routine statistics and medical registries

Clinical data (report of new cases and follow-up reports): CP Classification; Perinatal history; Diagnosis information; Possible CP causes; Neuroradiological examinations; Classification of motor skills (mobility, manual ability); Comorbidities, e.g. epilepsy, visual impairment, pain; Development and learning difficulties; Communication and nutrition; Hip and spinal pathologies (e.g. scoliosis); Treatments and therapies e.g. physiotherapy, hip surgery, medication; Socio-economic resources of the family.

Questionnaire data: Personal information; Health-related quality of life; Participation in daily life; Medical care and medication; Communication and dietary problems; Comorbidities; Treatments; Aids; Education and social environment; Family needs

Routine data and linkages: Communities; Federal Statistical Office (e.g. the birth register, cause of death statistics, hospital statistics); SwissNeoNet (register for premature and at-risk children).

Current status: From 2017-2021, the investigators have included 580 persons diagnosed with CP (Status May 31 2021; from birth year 1998)

The Swiss-CP-Reg contact new diagnosed persons with CP at regular intervals, and continuously analyse and publish data and findings.

Funding: Swiss Cerebral Foundation, Anna Mueller Grocholski Foundation, Swiss Academy of Childhood Disability SACD, Hand in Hand Anstalt, Ostschweizer Kinderspital and ACCENTUS Charitable Foundation (Walter Muggli Fund).

ELIGIBILITY:
Inclusion Criteria:

* Who were diagnosed with CP, confirmation of the diagnosis at the age of 5 years is required
* Who are born, treated for CP or living in Switzerland, and
* Who gave informed consent

Exclusion Criteria:

* Pure muscular hypotonia
* Neurometabolic diseases (e.g. neuronal storage diseases, leukodystrophies)
* Other progressive neurological diseases (e.g. spinocerebellar ataxias, hereditary spastic paraplegia, Rett syndrome, epileptic encephalopathy)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals living, born, or treated with a diagnosis of cerebral palsy in Switzerland
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2071-01 (Estimated); Study Completion 2071-01 (Estimated)

PRIMARY OUTCOMES:
Personal data | At diagnosis (age 0-5 years)
  Registering patients personal data
Change in date of registration | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in date of last consultation at physician for data collection
Birth history neonatal care | At diagnosis (age 0-5 years)
  Maternal birth history
Cause of change in vital status | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  what caused a change in patients vital status
Neonatal care | At diagnosis (age 0-5 years)
  Neonatal care
Age | At diagnosis (age 0-5 years)
  Age at diagnosis
Change in classification of CP | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in CP classification according to SCPE decision tree
Change in gross motor function | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of gross motor function
Change in fine motor function | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of fine motor function
Postneonatal CP | At diagnosis (age 0-5 years)
  Classification of postneonatal CP
Change in associated syndromes | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of associated syndromes using ICD code
Change of congenital anomalies | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of congenital anomalies using ICD code
Change of brain malformation | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of brain malformation using ICD code
Change in genetic syndromes | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in analysis results on genetic mutation
Change in neuroimaging | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration of change in neuro images
Change in anthropometrics | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration of change in anthropometric data
Change in sensory difficulties | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration of change in sensory capability
Change in nutrition | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration of change in feeding habits
Change in speech | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of verbal communication using VSS
Change in communication | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Change in classification of communication using CFCS
Change in comorbidities | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration of change in comorbidities
Change of hip | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Hip surveillance: registration of change in hip-dislocation
Change of scoliosis | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Assessing change in scoliosis using Cobb Winkel
Change in surgery | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in surgery history
Change in treatments | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in treatments
Change in therapies | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in therapies
Changes in medical equipment | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in use of medical equipment
Change in ancillary service | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in use of ancillary service
Change in mobility | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in mobility
Changes in behavior | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Assessing changes in behavior using scales
Changes in academic info | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in info on academic education
Changes in family history | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in info on health of family members
Changes in socio economics | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registering changes in info on parents socio-economic background
Changes in epilepsy | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Registration changes in epilepsy
Questionnaire data | 5-80 years
  Questionnaires focusing on specific research questions (Perinatal history, health related questions, health behavior, quality of life, participation, needs, concerns)
Change in cognition | follow-up data collection at regular intervals (at age of 5, 10 and 15 years, and at the time of transition to adult care (18±2 years))
  Assessing changes in mental ability using tests and school typ

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof. MD, Principal Investigator — Institute of Social and Preventive Medicine (ISPM), University of Bern
Locations (8):
- Switzerland (8):
  - University Children's Hospital Basel, UKBB, Basel
  - Pediatric Institute of Southern Switzerland, Ospedale San Giovanni, Bellinzona
  - Institute of Social and Preventive Medicine (ISPM), University of Bern, Bern
  - University Children's Hospital Bern, Inselspital, Bern
  - University Hospitals of Geneva, Geneva
  - University Children's hospital Lausane, CHUV, Lausanne
  - Children's Hospital of Eastern Switzerland, Sankt Gallen
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Researchers who wish to develop a nested study need to submit a proposal to the Swiss-CP-Reg committee and request permission. A concept sheet describing the planned analyses must be approved by the Swiss-CP-Reg committee. Nested studies might need separate ethics permission.

REFERENCES:
- [Result] Belle FN, Hunziker S, Fluss J, Grunt S, Juenemann S, Kuenzle C, Meyer-Heim A, Newman CJ, Ramelli GP, Weber P, Claudia E K, Tscherter A. Cohort profile: the Swiss Cerebral Palsy Registry (Swiss-CP-Reg) cohort study. Swiss Med Wkly. 2022 Feb 21;152:w30139. doi: 10.4414/smw.2022.w30139. eCollection 2022 Feb 14. PMID 35230014
- See also: Website of the registry — https://www.swiss-cp-reg.ch/